CLINICAL TRIAL: NCT00677729
Title: Inhaled Hypertonic Saline to Reduce Hospital Admissions in Infants With Viral Bronchiolitis (HS in ER Study)
Brief Title: Hypertonic Saline to Reduce Hospital Admissions in Bronchiolitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Queen's University (Other)
Collaborators: Kingston Health Sciences Centre (Other); Religious Hospitallers of Saint Joseph of the Hotel Dieu of Kingston (Unknown); Royal Victoria Hospital Of Barrie (Unknown)
Responsible Party: Principal Investigator, Dr. Michael Flavin, Principal Investigator, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSERFLA; PAED-214-08
Record Dates: First submitted 2008-05-02; First posted 2008-05-14 (Estimated); Last update posted 2015-11-13 (Estimated); Status verified 2015-11

CONDITIONS: Viral Bronchiolitis
Keywords: bronchiolitis; hypertonic saline; infants
MeSH Terms: conditions — Bronchiolitis, Viral; Bronchiolitis | interventions — Albuterol; Saline Solution, Hypertonic; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 4 ml of nebulized study solution containing 1 mg salbutamol plus 3% hypertonic saline (NaCl)
  Interventions: Drug: solution contains 1 mg salbutamol plus 3% hypertonic saline
- 2 (Placebo Comparator): 4 ml of nebulized study solution containing 1 mg salbutamol plus 0.9% saline (NaCl)
  Interventions: Drug: solution contains 1 mg salbutamol plus 0.9% saline

INTERVENTIONS:
Drug: solution contains 1 mg salbutamol plus 3% hypertonic saline — 4 ml of nebulized study solution containing 1 mg salbutamol plus 3% hypertonic saline every 20 minutes for a total of 3 doses
  Arms: 1
Drug: solution contains 1 mg salbutamol plus 0.9% saline — 4 ml of nebulized study solution containing 1 mg salbutamol plus 0.9% saline (NaCl) every 20 minutes for a total of 3 doses
  Arms: 2

SUMMARY:
Inhaled 3% hypertonic saline (HS) administered every 2-8 hours to infants admitted to hospital with viral bronchiolitis has been shown to improve airway clearance and reduces length of stay.

Hypothesis: When infants first present to the ER, frequent administration of HS over a brief time period will provide significant symptom improvement such that the need for hospital admission will be reduced.

Objective: To determine in a randomized, controlled and double-blind fashion if the short term intensive use of inhaled 3% hypertonic saline (HS) in the Emergency Room (ER) can reduce the rate of hospital admission for infants presenting with moderately severe viral bronchiolitis.

DETAILED DESCRIPTION:
Patients presenting to the Emergency Room (ER) or out-patient department with a diagnosis of moderately severe bronchiolitis (as defined by inclusion/exclusion criteria below) will be approached for entry into the study. After the initial routine assessment by the ER medical and nursing staff, informed consent will be obtained and the infant will be randomized to receive treatment in a double-blinded fashion with 4 ml of nebulized study solution containing 1 mg salbutamol (bronchodilator) plus either 3% hypertonic saline (HS, study group) or 0.9% saline (NS, control group) every 20 minutes for a total of 3 doses. After an observation period of 1 hour following the last dose, the infant will be reassessed by the attending physician in the ER for disposition (admit, discharge home, remain in ER for further treatment) at which point the infant's active involvement in the study will end. All subsequent therapy, if needed, will be at the sole discretion of the attending physician. The family of each recruited subject will be contacted by phone 7 days later to assess resolution of symptoms or the presence of any unexpected adverse effects.

Clinical response to the above treatment will also be determined independently by the study physician or designate utilizing a standardized respiratory scoring system, the Respiratory Distress Assessment Instrument (RDAI), at study entry and after the post-treatment observation period. The primary outcome measure is to compare the rate of admission to hospital between the study and control groups. A secondary outcome measure will involve the assessment of change in the RDAI between study entry and post-treatment.

The infant will remain in the ER throughout the study period and receive standard ongoing monitoring by the nursing staff. In the unlikely event of significant clinical worsening during this period, the ER physician on duty will be notified to assess and intervene as he/she feels appropriate. The site study investigator will be immediately notified of all such occurrences by the research assistant involved.

The study will be conducted over a single bronchiolitis season from November 1, 2008 to April 1, 2009. There will be 2 study sites as listed below with the name of the study site director.

* Royal Victoria Hospital of Barrie (Emergency Department), Barrie ON (B.A. Kuzik, MD, FRCP (lead investigator))
* Kingston General Hospital (Emergency Department) and Hotel Dieu Hospital (Emergency Department, Children's Outpatient Centre), Kingston ON (M. P. Flavin, MB, MRCP, FRCP)

ELIGIBILITY:
Inclusion Criteria:

1. < 24 months.
2. presenting to ER or outpatient department with moderately severe viral bronchiolitis defined as:

   1. history of viral upper respiratory tract infection within previous 7 days, plus
   2. presence of wheezing and/or crackles on chest auscultation, plus
   3. Respiratory Distress Assessment Instrument (RDAI, appendix B) score > 4 (of 17) or transcutaneous oxygen saturation (SaO2) < 94% in room air.

Patient exclusion criteria:

1. history of immunodeficiency or chronic cardiopulmonary disease (other than past history of wheezing).
2. critical illness at presentation.
3. use of nebulized HS within previous 12 hr.
4. prematurity (gestational age < 34 weeks).

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 81 (Actual)
Dates: Start 2008-11; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
compare the rate of admission to hospital between the study and control groups | 1 hour after treatment ends

SECONDARY OUTCOMES:
change in the RDAI between study entry and post-treatment. | 1 hour after treatment ends

CONTACTS AND LOCATIONS:
Overall Officials: Brian Kuzik, MD, Principal Investigator — The Royal Victoria Hospital of Barrie
Locations (3):
- Canada (3):
  - The Royal Victoria Hospital, Barrie, Ontario
  - Kingston General Hospital, Kingston, Ontario
  - Religious Hospitallers of Saint Joseph of the Hotel Dieu of Kingston, Kingston, Ontario

REFERENCES:
- [Derived] Kuzik BA, Flavin MP, Kent S, Zielinski D, Kwan CW, Adeleye A, Vegsund BC, Rossi C. Effect of inhaled hypertonic saline on hospital admission rate in children with viral bronchiolitis: a randomized trial. CJEM. 2010 Nov;12(6):477-84. doi: 10.1017/s1481803500012690. PMID 21073773